CLINICAL TRIAL: NCT06779656
Title: Regional Anesthesia Techniques in Breast Surgery: a Comparative Study
Brief Title: Regional Anesthesia Techniques in Breast Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-320
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Augmentation; Fibroadenoma; Mastectomy
MeSH Terms: conditions — Fibroadenoma | interventions — Anesthesia, General; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Paravertebral Block (PVB) (Experimental): The patient will be positioned in the lateral decubitus position with the operative side up. A high-frequency ultrasound probe (6-13 MHz) will be used to visualize the transverse processes, ribs, and pleura adjacent to the thoracic transverse processes on the operative side. Under ultrasound guidance, a needle will be inserted from posterior to anterior, advancing just superior to the tip of the transverse process, 1-2 mm, avoiding the pleura, and entering the paravertebral space. For ropivacaine, either 0.375% or 0.5% will be administered at a dose of 3-5 mL per segment, according to the patient's height and the extent of surgery. The block will target the T2-T6 nerve distribution, with a total dose not exceeding 20 mL. Alternatively, for liposomal bupivacaine (10-26.6 mg/mL), the dose will be determined based on the patient's weight and surgical extent, typically a total dose of 100-200 mg, diluted with normal saline to a total injection volume of 10-20 mL.
  Interventions: Device: General Anesthesia (GA); Procedure: Paravertebral Block (PVB)
- Rhomboid Intercostal and Subserratus Plane Block (RISS) (Experimental): The patient will be positioned in the lateral decubitus position with the operative side up. A high-frequency ultrasound probe will be used to locate the medial border of the scapula and identify the rhomboid, intercostal, and serratus anterior muscles. Under ultrasound guidance, the needle will be advanced into the plane between the rhomboid and intercostal muscles, or the plane between the intercostal and serratus anterior muscles. Ropivacaine 0.25% will be administered with an injection volume of 15-20 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 15-20 mL.
  Interventions: Device: General Anesthesia (GA); Procedure: Rhomboid Intercostal and Subserratus Plane Block (RISS)
- Pectoral Nerves Block II (PECS II) (Experimental): The patient will be placed in the supine position with the operative side arm slightly abducted. A high-frequency ultrasound probe will be used to locate the pectoralis major, pectoralis minor, and serratus anterior muscles. Under ultrasound guidance, the needle will be advanced into the plane between the pectoralis minor and serratus anterior muscles. Ropivacaine 0.25% will be administered with an injection volume of 20-30 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 20-30 mL.
  Interventions: Device: General Anesthesia (GA); Procedure: Pectoral Nerves Block II (PECS II)
- Intercostal Nerve Block (INB) (Experimental): The patient will be positioned in the lateral decubitus or supine position. A high-frequency ultrasound probe will be used to locate the ribs and intercostal muscles. Under ultrasound guidance, the needle will be advanced to the inferior margin of the rib, in the intercostal muscle plane. Ropivacaine 0.25% will be administered at a dose of 2-5 mL per intercostal space, typically targeting 3-5 intercostal spaces. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered at a dose of 2-5 mL per intercostal space, with a total dose not exceeding 200 mg, and a total injection volume of 5-20 mL.
  Interventions: Device: General Anesthesia (GA); Procedure: Intercostal Nerve Block (INB)
- Serratus Anterior Plane Block (SAPB) (Experimental): The patient will be positioned in the lateral decubitus or supine position with the operative side arm slightly abducted. A high-frequency ultrasound probe will be used to locate the serratus anterior muscle. Under ultrasound guidance, the needle will be advanced either superficial or deep to the serratus anterior muscle. Ropivacaine 0.25% will be administered with an injection volume of 20-30 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 20-30 mL.
  Interventions: Device: General Anesthesia (GA); Procedure: Serratus Anterior Plane Block (SAPB)
- Epidural Block (Experimental): The patient will be positioned in the sitting or lateral decubitus position. The area will be prepped and draped using standard aseptic technique. Either the thoracic or lumbar region will be selected, with the T4-T5 level often chosen. An epidural needle will be inserted into the epidural space, and an epidural catheter will be placed, using standard epidural techniques. Ropivacaine 0.1% or 0.083% will be administered as an initial bolus of 5-10 mL, followed by a continuous infusion at a rate of 5-10 mL/h. Alternatively, bupivacaine 0.1% or 0.0625% will be administered as an initial bolus of 5-10 mL, followed by a continuous infusion at a rate of 5-10 mL/h. These can be used in combination with opioid medications such as fentanyl or sufentanil to enhance analgesia.
  Interventions: Device: General Anesthesia (GA); Procedure: Epidural Block

INTERVENTIONS:
Device: General Anesthesia (GA) — Following administration of the regional anesthesia, general anesthesia with endotracheal intubation will be performed. Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.
Procedure: Paravertebral Block (PVB) — The patient will be positioned in the lateral decubitus position with the operative side up. A high-frequency ultrasound probe (6-13 MHz) will be used to visualize the transverse processes, ribs, and pleura adjacent to the thoracic transverse processes on the operative side. Under ultrasound guidance, a needle will be inserted from posterior to anterior, advancing just superior to the tip of the transverse process, 1-2 mm, avoiding the pleura, and entering the paravertebral space. For ropivacaine, either 0.375% or 0.5% will be administered at a dose of 3-5 mL per segment, according to the patient's height and the extent of surgery. The block will target the T2-T6 nerve distribution, with a total dose not exceeding 20 mL. Alternatively, for liposomal bupivacaine (10-26.6 mg/mL), the dose will be determined based on the patient's weight and surgical extent, typically a total dose of 100-200 mg, diluted with normal saline to a total injection volume of 10-20 mL.
  Arms: Paravertebral Block (PVB)
Procedure: Rhomboid Intercostal and Subserratus Plane Block (RISS) — The patient will be positioned in the lateral decubitus position with the operative side up. A high-frequency ultrasound probe will be used to locate the medial border of the scapula and identify the rhomboid, intercostal, and serratus anterior muscles. Under ultrasound guidance, the needle will be advanced into the plane between the rhomboid and intercostal muscles, or the plane between the intercostal and serratus anterior muscles. Ropivacaine 0.25% will be administered with an injection volume of 15-20 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 15-20 mL.
  Arms: Rhomboid Intercostal and Subserratus Plane Block (RISS)
Procedure: Pectoral Nerves Block II (PECS II) — The patient will be placed in the supine position with the operative side arm slightly abducted. A high-frequency ultrasound probe will be used to locate the pectoralis major, pectoralis minor, and serratus anterior muscles. Under ultrasound guidance, the needle will be advanced into the plane between the pectoralis minor and serratus anterior muscles. Ropivacaine 0.25% will be administered with an injection volume of 20-30 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 20-30 mL.
  Arms: Pectoral Nerves Block II (PECS II)
Procedure: Intercostal Nerve Block (INB) — The patient will be positioned in the lateral decubitus or supine position. A high-frequency ultrasound probe will be used to locate the ribs and intercostal muscles. Under ultrasound guidance, the needle will be advanced to the inferior margin of the rib, in the intercostal muscle plane. Ropivacaine 0.25% will be administered at a dose of 2-5 mL per intercostal space, typically targeting 3-5 intercostal spaces. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered at a dose of 2-5 mL per intercostal space, with a total dose not exceeding 200 mg, and a total injection volume of 5-20 mL.
  Arms: Intercostal Nerve Block (INB)
Procedure: Serratus Anterior Plane Block (SAPB) — The patient will be positioned in the lateral decubitus or supine position with the operative side arm slightly abducted. A high-frequency ultrasound probe will be used to locate the serratus anterior muscle. Under ultrasound guidance, the needle will be advanced either superficial or deep to the serratus anterior muscle. Ropivacaine 0.25% will be administered with an injection volume of 20-30 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 20-30 mL.
  Arms: Serratus Anterior Plane Block (SAPB)
Procedure: Epidural Block — The patient will be positioned in the sitting or lateral decubitus position. The area will be prepped and draped using standard aseptic technique. Either the thoracic or lumbar region will be selected, with the T4-T5 level often chosen. An epidural needle will be inserted into the epidural space, and an epidural catheter will be placed, using standard epidural techniques. Ropivacaine 0.1% or 0.083% will be administered as an initial bolus of 5-10 mL, followed by a continuous infusion at a rate of 5-10 mL/h. Alternatively, bupivacaine 0.1% or 0.0625% will be administered as an initial bolus of 5-10 mL, followed by a continuous infusion at a rate of 5-10 mL/h. These can be used in combination with opioid medications such as fentanyl or sufentanil to enhance analgesia.
  Arms: Epidural Block

SUMMARY:
This clinical trial aims to evaluate the efficacy of liposomal bupivacaine and ropivacaine, when administered via paravertebral block, the rhomboid intercostal and subserratus plane (RISS) block, PECS II block, intercostal nerve block, serratus anterior plane block, or epidural block, in patients undergoing breast surgery (including augmentation, fibroadenoma excision, and mastectomy). The primary objectives are to determine:

1. Whether the use of liposomal bupivacaine or ropivacaine reduces the postoperative analgesic requirements in participants.
2. What potential adverse events participants experience when using liposomal bupivacaine or ropivacaine.
3. Which of the following regional anesthesia techniques provides superior analgesia: paravertebral block, RISS block, PECS II block, intercostal nerve block, serratus anterior plane block, or epidural block.

Participants will undergo one of the following regional anesthesia techniques upon arrival to the surgical suite: paravertebral block, RISS block, PECS II block, intercostal nerve block, serratus anterior plane block, or epidural block. Following regional anesthesia administration, general anesthesia with endotracheal intubation will be performed. Participants' vital signs, postoperative analgesic consumption, and recovery will be recorded.

DETAILED DESCRIPTION:
Study design：This study is a prospective, randomized, comparative, blinded clinical trial, evaluating both superiority and non-inferiority. The study will compare the analgesic efficacy of paravertebral block, the rhomboid intercostal and subserratus plane (RISS) block, PECS II block, intercostal nerve block, serratus anterior plane block, and epidural block for breast surgery (including augmentation, fibroadenoma excision, and mastectomy). Participants and clinician blinding will be implemented. Patient recruitment will take place at Baogang Hospital in Inner Mongolia. This study was approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia and adhered to the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed consent voluntarily.

Patients: This study will enroll 180 patients, ASA physical status I-III, aged 18 years or older, scheduled for breast surgery (including augmentation, fibroadenoma excision, and mastectomy) between February and May 2025. Participants will be randomly assigned to one of six groups: paravertebral block, rhomboid intercostal and subserratus plane (RISS) block, PECS II block, intercostal nerve block, serratus anterior plane block, or epidural block, with 30 patients in each group.

Randomization and Blinding: Block randomization was used to generate the random allocation sequence. A block size of 6 was utilized, and the random sequence was generated using the 'blockrand' package in R version 4.3.2. An independent third party performed the allocation of the random sequence. Allocation concealment was ensured using sequentially numbered, sealed, opaque envelopes. The research team was blinded throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention: Upon arrival to the operating room, participants will be monitored with electrocardiography, blood pressure, and pulse oximetry. Participants will be placed in the prone position with their arms abducted and internally rotated. Ultrasound guidance will be used for all regional anesthesia procedures (SonoSite Edge II; Fujifilm SonoSite, Bothell, WA, USA) with a linear 13-6 MHz ultrasound probe (HFL50x; Fujifilm SonoSite, Bothell, WA, USA). For each block, a 5 mL test dose will be injected initially, followed by observation for clinical signs of a successful block. After confirming correct placement, the remaining dose of the anesthetic agent will be injected. Following administration of the regional anesthesia, general anesthesia with endotracheal intubation will be performed. Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.

1. Paravertebral Block (PVB) The participant will be positioned in the lateral decubitus position with the operative side up. A high-frequency ultrasound probe (6-13 MHz) will be used to visualize the transverse processes, ribs, and pleura adjacent to the thoracic transverse processes on the operative side. Under ultrasound guidance, a needle will be inserted from posterior to anterior, advancing just superior to the tip of the transverse process, 1-2 mm, avoiding the pleura, and entering the paravertebral space. For ropivacaine, either 0.375% or 0.5% will be administered at a dose of 3-5 mL per segment, according to the patient's height and the extent of surgery. The block will target the T2-T6 nerve distribution, with a total dose not exceeding 20 mL. Alternatively, for liposomal bupivacaine (10-26.6 mg/mL), the dose will be determined based on the patient's weight and surgical extent, typically a total dose of 100-200 mg, diluted with normal saline to a total injection volume of 10-20 mL.
2. Rhomboid Intercostal and Subserratus Plane Block (RISS) The participant will be positioned in the lateral decubitus position with the operative side up. A high-frequency ultrasound probe will be used to locate the medial border of the scapula and identify the rhomboid, intercostal, and serratus anterior muscles. Under ultrasound guidance, the needle will be advanced into the plane between the rhomboid and intercostal muscles, or the plane between the intercostal and serratus anterior muscles. Ropivacaine 0.25% will be administered with an injection volume of 15-20 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 15-20 mL.
3. Pectoral Nerves Block II (PECS II) The participant will be placed in the supine position with the operative side arm slightly abducted. A high-frequency ultrasound probe will be used to locate the pectoralis major, pectoralis minor, and serratus anterior muscles. Under ultrasound guidance, the needle will be advanced into the plane between the pectoralis minor and serratus anterior muscles. Ropivacaine 0.25% will be administered with an injection volume of 20-30 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 20-30 mL.
4. Intercostal Nerve Block (INB) The participant will be positioned in the lateral decubitus or supine position. A high-frequency ultrasound probe will be used to locate the ribs and intercostal muscles. Under ultrasound guidance, the needle will be advanced to the inferior margin of the rib, in the intercostal muscle plane. Ropivacaine 0.25% will be administered at a dose of 2-5 mL per intercostal space, typically targeting 3-5 intercostal spaces. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered at a dose of 2-5 mL per intercostal space, with a total dose not exceeding 200 mg, and a total injection volume of 5-20 mL.
5. Serratus Anterior Plane Block (SAPB) The participant will be positioned in the lateral decubitus or supine position with the operative side arm slightly abducted. A high-frequency ultrasound probe will be used to locate the serratus anterior muscle. Under ultrasound guidance, the needle will be advanced either superficial or deep to the serratus anterior muscle. Ropivacaine 0.25% will be administered with an injection volume of 20-30 mL. Alternatively, liposomal bupivacaine (10-26.6 mg/mL) will be administered according to the manufacturer's recommended dosage, usually a total dose of 100-200 mg, with an injection volume of 20-30 mL.
6. Epidural Block The participant will be positioned in the sitting or lateral decubitus position. The area will be prepped and draped using standard aseptic technique. Either the thoracic or lumbar region will be selected, with the T4-T5 level often chosen. An epidural needle will be inserted into the epidural space, and an epidural catheter will be placed, using standard epidural techniques. Ropivacaine 0.1% or 0.083% will be administered as an initial bolus of 5-10 mL, followed by a continuous infusion at a rate of 5-10 mL/h. Alternatively, bupivacaine 0.1% or 0.0625% will be administered as an initial bolus of 5-10 mL, followed by a continuous infusion at a rate of 5-10 mL/h. These can be used in combination with opioid medications such as fentanyl or sufentanil to enhance analgesia.

Outcomes and Measures: Patient follow-up will be conducted in the hospital ward by two specifically trained nurses, who will be blinded to patient allocation. Assessments will occur at four time points: before therapy (baseline), on the day of therapy (Day 1), and on Day 7 post-therapy. These assessments will be performed either in person or via telephone.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification I-III.
* Age of 18 years or older.
* Scheduled to undergo breast surgery, including augmentation, fibroadenoma excision, or mastectomy.

Exclusion Criteria:

* Known allergy to local anesthetics.
* Pregnancy or lactation.
* Coagulation disorders.
* Severe cardiopulmonary disease.
* Local infection at the injection site.
* Unstable psychiatric illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | At baseline (before therapy),At 2hours post-surgery, At 6hours post-surgery、At 12hours post-surgery、At 24hours post-surgery.
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.
Total Analgesic Consumption within 24 Hours Post-Surgery | At baseline (in operation),At 2hours post-surgery, At 6hours post-surgery、At 12hours post-surgery、At 24hours post-surgery.
  The total amount of all analgesic medications (including opioids such as fentanyl and morphine, and non-steroidal anti-inflammatory drugs such as ibuprofen and acetaminophen) used by the patient within the first 24 hours following surgery will be recorded. These dosages will be converted to their equivalent morphine milligram (mg) dose. Higher total morphine equivalent doses will indicate a lower level of analgesia efficacy.

SECONDARY OUTCOMES:
Patient Satisfaction Score | At 24 hours post-surgery
  Patient satisfaction with postoperative analgesia will be assessed using a patient satisfaction questionnaire. The questionnaire utilizes a 10-point numerical rating scale, where 0 represents "completely dissatisfied" and 10 represents "extremely satisfied." The questionnaire will include evaluations of pain control, comfort, and trust in the medical team.
Postoperative Recovery Status | Assessments will be performed at 6 hours, 12 hours, and 24 hours post-surgery, with a final assessment prior to hospital discharge.
  The Modified Postoperative Recovery Score (mPORAS) will be used to assess postoperative recovery status, including physiological recovery, pain control, mobility, and psychological state. Each item will be scored on a scale of 0 to 4, with a total score ranging from 0 to 20. Higher scores will indicate better postoperative recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2031
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.